CLINICAL TRIAL: NCT02746666
Title: Influence of a Clinical Pharmacist's Intervention on Quality of Life of a Breast Cancer Patient Under Adjuvant Chemotherapy
Brief Title: Pharmacist's Influence on Breast Cancer Patient Quality of Life
Acronym: PIBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Sestre Milosrdnice (Other)
Responsible Party: Principal Investigator, Robert Šeparović, MD PHD, University Hospital Sestre Milosrdnice
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1705201504032016
Record Dates: First submitted 2016-04-09; First posted 2016-04-21 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer, Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Under pharmacist's behavioral intervention
  Interventions: Behavioral: Pharmacist's behavioral intervention
- Control (No Intervention): No pharmacist's behavioral intervention

INTERVENTIONS:
Behavioral: Pharmacist's behavioral intervention — Pharmacist's 30 min counselling on antiemetic therapy, causes of nausea or vomiting and ways to prevent them during chemotherapy.
  Arms: Intervention

SUMMARY:
The purpose of this study is to investigate the impact of pharmacist behavioral intervention's influence on breast cancer patients' quality of life. Croatian randomized controlled trial. Targeted population: general population of breast cancer patients under the first adjuvant anthracycline chemotherapy. Primary outcome: difference in EORTC QLQ-BR23 questionnaire result from the baseline to after 3 week cycle.

ELIGIBILITY:
Inclusion Criteria:

* Early breast cancer
* First adjuvant chemotherapy
* Chemotherapy protocol: anthracycline x 4

Exclusion Criteria:

* Cardiovascular comorbidities
* Regular nausea or vomiting during six months before enrollment
* Unable to answer the quality of life questionnaire on their own

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
changes in quality of life of a breast cancer patient under chemotherapy, after a clinical pharmacist's behavioral intervention, measured by EORTC B23 questionnaire | up to two months